CLINICAL TRIAL: NCT04049006
Title: Primary Care as a Promoter of the Quality of Life of Fibromyalgia Patients. Effectiveness and Cost-utility of a Complex Intervention Through a Randomized Clinical Trial
Brief Title: Effectiveness and Cost-utility of a Complex Intervention for Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PI1800943
Record Dates: First submitted 2019-05-22; First posted 2019-08-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2019-08

CONDITIONS: Fibromyalgia
Keywords: Quality of life; randomized Controlled trials; Costs and Cost analysis; Primary Health Care
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- complex-treatment benefiting group (Experimental): Participants in the intervention group will receive the complex treatment and the usual clinical practice.
  Interventions: Other: complex treatment
- complex-treatment no benefiting group (No Intervention): Participants in the control group will receive the care from the usual clinical practice

INTERVENTIONS:
Other: complex treatment — The complex treatment will be based on health education, aerobic physical exercise and cognitive-behavioral therapy, during 12 weeks in sessions of 2 hours/week. The sessions will be conducted in the primary health care by trained professionals.
  Arms: complex-treatment benefiting group

SUMMARY:
Fibromyalgia (FM) is a chronic disease characterized by chronic pain, fatigue and loss of function that leads to a significant deterioration in the quality of life. Despite controversies about the most appropriate treatment, studies indicate that a multidisciplinary treatment would be effective. This study aims to analyze the effectiveness and cost-utility of a complex intervention in the quality of life (main variable), the functional impact, the mood and the pain of people with FM treated in the Primary Care Teams (PCTs) of the Catalan Institute of Health (CIH).

DETAILED DESCRIPTION:
Methods and analysis: Mixed methodology study following the recommendations of the Medical Research Council, with two phases. Phase 1: Randomized pragmatic clinical trial with patients diagnosed with FM and assigned to one of the 11 PCTs of the CIH (Territorial management of "Terras del Ebro"). A total sample of 336 patients is estimated.

The usual clinical practice will be carried out in the control group and the usual practice and the complex treatment, in the intervention group. The complex treatment will be based on health education, aerobic physical exercise and cognitive-behavioral therapy, during 12 weeks in sessions of 2 hours/week. Statistical analysis: Assessment of the standardized mean response and of the size of the standardized effect and multivariate logistic regression analysis will be performed. The economic analysis will be based on useful measures. Phase 2: Qualitative socio-constructivist study to identify the improvement aspects of the intervention according to the results obtained and the opinions and experiences of the participants (patients and professionals). The sampling will be theoretical with 2 discussion groups composed of participants in the intervention and 2 discussion groups of professionals from different PCTs.

ELIGIBILITY:
Inclusion Criteria (all criteria must be met):

* Have a clinical diagnosis of fibromyalgia
* Have a fixed or mobile telephone
* Voluntarily accept participation in the project

Exclusion Criteria:

* Active psychotic outbreak;
* Intellectual deficiency;
* Severe depression and personality disorder;
* Self and hetero-aggressive behaviors;
* Individual assessment of active consumption of psychoactive substances;
* Incompatibility with the group's schedule.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in life quality | change from life quality at 3, 9 and 15 months after the beginning of the study
  to be evaluated with the health questionnaire (SF-36v2). It will be measured by a scale Likert: 0 (worst) to 100 (best).
Change in functional impact of fibromyalgia | Change from functional impact of fibromyalgia at 3, 9 and 15 months after the beginning of the study.
  to be evaluated with the Revised Questionnaire on the Impact of Fibromyalgia (FIQR) It will be measured by a scale Likert: 0 (best) to 100 (worst).
Change in tender points | Change from tender points at 3, 9 and 15 months after the beginning of the study.
  Tender points evaluate the presence of pain in 18 areas of the body and will be measured by a scale Likert: 0 (best) to 18 (worst).
Change in Visual Analog Scale for pain (VAS) | Change from VAS at 3, 9 and 15 months after the beginning of the study.
  The VAS evaluates the self-perceived intensity of pain by a scale Likert: 0 (absence of pain) to 10 (worst possible pain).
Change in mood indicator (anxiety) | Change from mood indicator (anxiety) at 3, 9 and 15 months after the beginning of the study.
  To be evaluated with the Hospital Anxiety and Depression Scale (HADS) questionnaire. The scale likert punctuates from 0 to 21 (8 to 10 indicates a doubtful case of anxiety; more than 11 indicates a probable case of anxiety).
Change in mood indicator (depression) | Change from mood indicator (depression) at 3, 9 and 15 months after the beginning of the study.
  To be evaluated with the Hospital Anxiety and Depression Scale (HADS) questionnaire. The scale likert punctuates from 0 to 21 (8 to 10 indicates a doubtful case of anxiety; more than 11 indicates a probable case of anxiety).

SECONDARY OUTCOMES:
Sociodemographic characteristics of the patients | baseline (pre intervention period)
  age, sex, level of education, work disability and family coexistence
Presence/absence of physical manifestations | baseline (pre intervention period)
  Physical manifestations to be evaluated: non-repairing sleep, excessive fatigue, dryness of mucous membranes, Raynaud's phenomenon, Intolerance to olfactory and auditory stimuli, cephalgia lumbar, increased sensitivity to the side effects of drugs and paresthesia of hands and feet. To be evaluated with a questionnaire (yes/no type)
Presence/absence of physical or psychic trigger factor of fibromyalgia | baseline (pre intervention period)
  To be evaluated with a questionnaire (yes/no type)
Presence/absence of physical, psychic or psychological factor responsible for fibromyalgia maintenance | baseline (pre intervention period)
  To be evaluated with a questionnaire (yes/no type)
Presence/absence of family history of fibromyalgia | baseline (pre intervention period)
  To be evaluated with a questionnaire (yes/no type)
presence/absence of cognitive psychological symptoms: Difficulty for concentration, alteration of memory | baseline (pre intervention period)
  To be evaluated with a questionnaire (yes/no type)
presence/absence of comorbidities: Chronic pelvic pain, dysmenorrhoea, irritable bladder syndrome, myofascial pain | baseline (pre intervention period)
  To be evaluated with a questionnaire (yes/no type)
Diagnosis date | baseline (pre intervention period)
  diagnosis date of fibromyalgia
Years of evolution | baseline (pre intervention period)
  years of evolution of fibromyalgia
presence/absence of pathological history: arthrosis, arthritis and mental health problems | baseline (pre intervention period)
  To be evaluated with a questionnaire (yes/no type)
Test of the thyroid stimulating hormone | baseline (pre intervention period)
  Analytic results in milliunits per litre (mUI/L)
Hemogram | baseline (pre intervention period)
  Analytic results of hemogram
Glucose, creatinine and C-reactive protein tests | baseline (pre intervention period)
  Analytic results of each test in mg/dl
Liver Function Tests | baseline (pre intervention period)
  Analytic results of each test
Globular sedimentation rate | baseline (pre intervention period)
  Analytic results in mm
Rheumatoid factor | baseline (pre intervention period)
  Analytic results in IU/mL
Pharmacy billing cost | one year before the beginning of the intervention in comparison with one year after the beginning of the intervention
  antidepressants, analgesics and others
Cost of visits | one year before the beginning of the intervention in comparison with one year after the beginning of the intervention
  cost of visits to family doctor or nurse and cost of urgency visits
Cost of referrals | one year before the beginning of the intervention in comparison with one year after the beginning of the intervention
  cost of referrals to external consultations
Cost of lost productivity | one year before the beginning of the intervention in comparison with one year after the beginning of the intervention
  cost of lost productivity due to sick leave

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Català de la Salut, Tortosa, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Some individual participant data collected during the qualitative phase of the study, after deidentification, will be published in articles. Some articles were already published.
  Grouped (not individual) participant data that underlie the quantitative results of the trial (and also qualitative results) will be published in text, tables, or figures. The quantitative results were not yet published.
  Study protocols and patients' qualitative data of this project were already published.
Supporting Information: Study Protocol
Time Frame: The data will be available in the scientific publications derived from the project.
Access Criteria: Through scientific publications in open access journals

REFERENCES:
- [Result] Caballol Angelats R, Goncalves AQ, Aguilar Martin C, Sancho Sol MC, Gonzalez Serra G, Casajuana M, Carrasco-Querol N, Fernandez-Saez J, Dalmau Llorca MR, Abellana R, Berenguera A; SensiTEbre group. Effectiveness, cost-utility, and benefits of a multicomponent therapy to improve the quality of life of patients with fibromyalgia in primary care: A mixed methods study protocol. Medicine (Baltimore). 2019 Oct;98(41):e17289. doi: 10.1097/MD.0000000000017289. PMID 31593081
- [Result] Arfuch VM, Caballol Angelats R, Aguilar Martin C, Carrasco-Querol N, Sancho Sol MC, Gonzalez Serra G, Fuste Anguera I, Goncalves AQ, Berenguera A. Assessing the benefits on quality of life of a multicomponent intervention for fibromyalgia syndrome in primary care: patients' and health professionals' appraisals: a qualitative study protocol. BMJ Open. 2020 Nov 11;10(11):e039873. doi: 10.1136/bmjopen-2020-039873. PMID 33177139
- [Result] Arfuch VM, Aguilar Martin C, Berenguera A, Caballol Angelats R, Carrasco-Querol N, Gonzalez Serra G, Sancho Sol MC, Fuste Anguera I, Fernandez Saez J, Goncalves AQ, Casajuana M. Cost-utility analysis of a multicomponent intervention for fibromyalgia syndrome in primary care versus usual clinical practice: study protocol for an economic evaluation of a randomised control trial. BMJ Open. 2021 Feb 5;11(2):e043562. doi: 10.1136/bmjopen-2020-043562. PMID 33550259
- [Result] Arfuch VM, Queiroga Goncalves A, Caballol Angelats R, Aguilar Martin C, Carrasco-Querol N, Sancho Sol MC, Gonzalez Serra G, Fuste Anguera I, Berenguera A. Patients' appraisals about a multicomponent intervention for fibromyalgia syndrome in primary care: a focus group study. Int J Qual Stud Health Well-being. 2021 Dec;16(1):2005760. doi: 10.1080/17482631.2021.2005760. PMID 34839810
- [Result] Arfuch VM, Caballol Angelats R, Aguilar Martin C, Goncalves AQ, Carrasco-Querol N, Gonzalez Serra G, Sancho Sol MC, Fuste Anguera I, Friberg E, Berenguera A. Patients' Lived Experience in a Multicomponent Intervention for Fibromyalgia Syndrome in Primary Care: A Qualitative Interview Study. Int J Environ Res Public Health. 2022 Oct 15;19(20):13322. doi: 10.3390/ijerph192013322. PMID 36293900
- [Derived] Caballol Angelats R, Goncalves AQ, Abellana R, Carrasco-Querol N, Pamies Corts A, Gonzalez Serra G, Gracia Benaiges D, Sancho Sol MC, Fuste Anguera I, Chavarria Jordana S, Cuevas Baticon B, Batlle Escolies G, Fibla Reverte M, Espuny Valles N, Buera Pitarque N, Marti Cavalle M, Suazo NP, Estivill Bargallo J, Lopez Guerrero MA, Lopez Guerrero C, Perez Acin P, Matamoros Callarisa I, Baucells J, Suazo Ciurana A, Fernandez-Saez J, Dalmau Llorca MR, Berenguera A, Aguilar Martin C. Effectiveness of a Multicomponent Program for Fibromyalgia Patients in a Primary Care Setting (FIBROCARE Program): A Pragmatic Randomized Controlled Trial. J Clin Med. 2024 Dec 30;14(1):161. doi: 10.3390/jcm14010161. PMID 39797245
- [Derived] Arfuch VM, Aguilar Martin C, Berenguera A, Caballol Angelats R, Goncalves AQ, Carrasco-Querol N, Gonzalez Serra G, Sancho Sol MC, Fuste Anguera I, Friberg E, Pettersson E, Casajuana M. Cost-utility of a multicomponent intervention for fibromyalgia versus usual care: a pragmatic randomised controlled trial. J Rehabil Med. 2023 Dec 19;55:jrm12361. doi: 10.2340/jrm.v55.12361. PMID 38111994